CLINICAL TRIAL: NCT05727917
Title: Efficacy and Safety of Hetrombopag for the Enhancement of Platelet Engraftment After Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Hematological Disease
Brief Title: Hetrombopag for the Enhancement of Platelet Engraftment After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230131
Record Dates: First submitted 2023-02-06; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Hematological Disease; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Diseases | interventions — hetrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hetrombopag group (Experimental group) (Experimental): After hematopoietic stem cell reinfusion, the patients begin to take hetrombopag orally 7.5mg/d, until the patients reach complete platelet response (CR, platelet count ≥50×109/L for 3 consecutive days without platelet transfusions for 7 consecutive days). The treatment will stop when patients accept 21 consecutive days of treatment or reach the discontinuation criteria.
  Interventions: Drug: Hetrombopag
- Control group (Placebo Comparator): After hematopoietic stem cell transfusion, the patients will be only observed, and the observation during the treatment period will be ended after 30 days.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Hetrombopag — After hematopoietic stem cell reinfusion, the patients begin to take hetrombopag orally 7.5mg/d, until the patients reach complete platelet response.The treatment will stop when patients accept 21 consecutive days of treatment or reach the discontinuation criteria.
  Arms: hetrombopag group (Experimental group)
Other: placebo — After hematopoietic stem cell transfusion, the patients will be only observed, and the observation during the treatment period will be ended after 30 days
  Arms: Control group

SUMMARY:
This investigator-initiated, prospective, multicenter, open-label, randomized, controlled clinical study is designed to evaluate the clinical efficacy and safety of hetrombopag for promoting platelet engraftment after allo-HSCT in patients with hematological disease.

After signing the informed consent form, the patients will enter the screening period (up to 14 days), and the qualified patients will be randomly selected into the experimental group and the control group according to the ratio of 1:1.

Experimental group: After hematopoietic stem cell reinfusion, the patients begin to take hetrombopag orally 7.5mg/d, until the patients reach complete platelet response (CR, platelet count ≥ 50×109/L for 3 consecutive days without platelet transfusions for 7 consecutive days). The treatment will stop when patients accept 21 consecutive days of treatment or reach the discontinuation criteria.

Control group: After hematopoietic stem cell transfusion, the patients will be only observed, and the observation during the treatment period will be ended after 30 days.

Patients will continue to enter the follow-up period (+ 100 days after transplantation) and the survival follow-up period (1 year after transplantation) after the end of the treatment period.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective treatment for many hematological diseases. Thrombocytopenia is a common complication of allo-HSCT. Incidence ranged from 5% to 37%. In order to promote the transplantation of donor stem cells and reduce the incidence of graft versus host disease (GVHD) and disease recurrence, high-dose chemotherapy, radiotherapy and other pretreatment schemes are usually used before operation to induce immune tolerance and eliminate tumor cells to the greatest extent. At the same time, the recipient's bone marrow was in an "empty" state before the donor's stem cell engraftment. At this time, the hematopoietic function of the bone marrow was severely inhibited, and the blood cell count was very low. Generally, the platelet count was less than 20 × 10^9/L within 13-54 days. Patients whose time to platelet recovery ≥ 50 × 10^9/L was greater than 60 days had a significant increase in transplant-related mortality rate and a significant decrease in long-term survival. Therefore, it is very important to prevent and treat thrombocytopenia after hematopoietic stem cell transplantation.

To date, no standard treatment has been proposed for thrombocytopenia after allo-HSCT. In order to prevent bleeding, patients often need multiple platelet transfusions for a long time, which increases the economic burden, and platelet transfusion may also lead to many adverse reactions, such as anaphylactic shock, acute lung injury, heart failure, viral infection, etc. Some patients may also have ineffective platelet transfusion. In addition, prolonged blood transfusion consumes a lot of hospital resources and costs, and reduces the quality of life of patients. The 2021 edition of the Chinese Expert Consensus on the Management of Hemorrhagic Complications after Hematopoietic Stem Cell Transplantation suggests that patients with thrombocytopenia after transplantation should actively control the inducing factors. In addition to platelet transfusion, recombinant human thrombopoietin (rhTPO) 300 U/kg/d subcutaneous injection can be used, and TPO receptor agonists can also be tried. Platelet counts > 50 × 109/L1 were maintained.

Thrombopoietin (TPO) is the most important cytokine that promotes platelet production in humans. TPO promotes platelet production by binding to the TPO receptor (TPO-R) on the cell surface. TPO receptor agonist (TPO-RA) activates downstream STAT/MAPK signaling pathway by binding and activating TPO receptor, which effectively stimulates platelet production, increases platelet count and reduces the occurrence of bleeding events. At present, TPO-RA in clinical application includes recombinant human thrombopoietin (rhTPO), peptide TPO-RA (Romiplostim), non-peptide TPO RA (Hetrombopag, Eltrombopag, Avatrombopag, etc.), which is widely used in various thrombocytopenia, including primary immune thrombocytopenia (ITP). Aplastic anemia (AA), chemotherapy-induced thrombocytopenia (CIT) and perioperative thrombocytopenia in patients with liver diseases have good efficacy and safety. Han et al. conducted a prospective randomized controlled study to explore the role of rhTPO in promoting platelet engraftment after haplo-HSCT. The rhTPO group was given rhTPO 15000U subcutaneously once a day from the first day after transplantation. Discontinue when platelet count ≥ 50 × 109/L for more than 3 days; The incidence of platelet engraftment was significantly higher in the rhTPO group than in the control group on day + 60 after transplantation (91.7 ± 3.8% vs. 74.5 ± 5.8%, p = 0.041), and the number of platelet transfusions during + 14d to + 60d was significantly reduced (4 ± 5 vs. 7 ± 9, p = 0.018), suggesting that routine use of thrombopoiesis drugs after transplantation can effectively promote platelet engraftment and reduce the need for platelet transfusion therapy, which is a safe and effective treatment. Other TPO receptor agonists have been reported to be effective in the treatment of thrombocytopenia after hematopoietic stem cell transplantation, but there is no consensus on the optimal timing and dosage. With the continuous progress of transplantation technology in China, the indications of HSCT have been further broadened, the number of cases has continued to grow, and more clinical evidence is needed.

Hetrombopag is a new generation of oral small molecule non-peptide TPO-RA independently developed by Jiangsu Hengrui Pharmaceutical Co., Ltd. In June 2021, it was approved by NMPA for the treatment of adult chronic ITP patients who did not respond well to glucocorticoid, immunoglobulin and other treatments, as well as adult SAA patients who did not respond well to immunosuppressive therapy. Pharmacological studies at the protein level showed that the phosphorylation of various signaling proteins was significantly stronger at the same dose than that of eltrombopag. Compared with rhTPO, it has a more lasting and stable effect on the phosphorylation level of downstream signals. There is great potential for the clinical application of hetrombopag in hematopoietic stem cell transplantation, but the efficacy and safety of hetrombopag in promoting platelet engraftment after transplantation need to be further verified.

Thus,this investigator-initiated, prospective, multicenter, open-label, randomized, controlled clinical study is designed to evaluate the clinical efficacy and safety of hetrombopag for promoting platelet engraftment after allo-HSCT in patients with hematological disease.

After signing the informed consent form, the patients will enter the screening period (up to 14 days), and the qualified patients will be randomly selected into the experimental group and the control group according to the ratio of 1:1.

Experimental group: After hematopoietic stem cell reinfusion, the patients begin to take hetrombopag orally 7.5mg/d, until the patients reach complete platelet response (CR, platelet count ≥ 50×10^9/L for 3 consecutive days without platelet transfusions for 7 consecutive days). The treatment will stop when patients accept 21 consecutive days of treatment or reach the discontinuation criteria.

Control group: After hematopoietic stem cell transfusion, the patients will be only observed, and the observation during the treatment period will be ended after 30 days.

Patients will continue to enter the follow-up period (+ 100 days after transplantation) and the survival follow-up period (1 year after transplantation) after the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. The patients signed the informed consent and participated in the study voluntarily;
2. Age ≥ 18 years old, regardless of gender;
3. ECOG score ≤ 2;
4. Expected survival ≥ 3 months;
5. Patients with hematological diseases who received allo-HSCT for the first time;
6. The patient's laboratory tests met the following criteria:

   1. Alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN), Aspartate aminotransferase (AST) ≤ 3.0 × ULN;
   2. Serum total bilirubin ≤ 1.5 × ULN;
   3. Serum creatinine ≤ 1.5 × ULN;
7. Investigators evaluated that patients would benefit from hetrombopag.

Exclusion Criteria:

1. History of allergy to TPO-RA drugs;
2. Previous bone marrow or hematopoietic stem cell transplantation;
3. Hematologic malignancies did not reach complete remission before transplantation;
4. Central nervous system leukemia;
5. Arterial or venous thrombosis, such as cerebral infarction, pulmonary embolism, arterial thrombosis, deep venous thrombosis and disseminated intravascular coagulation (DIC), occurred within 6 months before the screening period;
6. Heart disease, such as New York Heart Association (NYHA) class III/IV congestive heart failure, angina pectoris, myocardial infarction, and arrhythmias requiring treatment, occurring within 6 months before the screening period;
7. Prolonged QT syndrome during the screening period;
8. Active hepatitis B or hepatitis C;
9. Positive for anti-HIV antibodies or anti-TP antibodies;
10. Active infection that is difficult to control;
11. Pregnant or breastfeeding women;
12. Other conditions not suitable for inclusion evaluated by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with platelet engraftment within 21 days after transplantation | 21 days after transplantation
  Proportion of patients who maintained platelet count ≥ 20 × 10^9/L without platelet transfusion for 7 consecutive days within 21 days after transplantation

SECONDARY OUTCOMES:
Median time to platelet engraftment | 100 days
  the first day when the platelet count ≥ 20 × 10^9/L for 7 consecutive days
Median time to neutrophil engraftment | 100 days
  the first day when the absolute neutrophil count ≥ 0.5 × 10^9/L for 3 consecutive days
Proportion of patients with neutrophil engraftment within 21 days after transplantation | 21 days after transplantation
  proportion of patients with absolute neutrophil count ≥ 0.5 × 10^9/L for 3 consecutive days within 21 days after transplantation
Proportion of patients with platelet engraftment within 30 days after transplantation | 30 days after transplantation
  proportion of patients who maintained platelet count ≥ 20 × 10^9/L without platelet transfusion for 7 consecutive days within 30 days after transplantation
Platelet complete response rate (CR) within 30 days after transplantation | 30 days after transplantation
  proportion of patients who maintained platelet count ≥ 50×10^9/L for 3 consecutive days without platelet transfusions for 7 consecutive days within 30 days after transplantation
Platelet transfusion volume | 100 days
  total platelet transfusion volume within 100 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Erlie Jiang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No